CLINICAL TRIAL: NCT07090083
Title: Pediatric MASLD and Food Insecurity
Brief Title: Pediatric Metabolic Dysfunction-associated Steatotic Liver Disease and Food Insecurity
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: American Gastroenterological Association Foundation (Other); UCSF Population Health Health Equity Award (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23-40614
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Food Insecurity
Keywords: MASLD; food insecurity; pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Food secure: Children with MASLD with exposure to household food security
- Food insecure: Children with MASLD with exposure to household food insecurity

SUMMARY:
This proposal addresses a critical gap in our understanding of the impact of household food insecurity (FI) on pediatric metabolic dysfunction-associated steatotic liver disease (MASLD) severity. There is evidence that children in families that do not have the ability to provide consistently healthy and high-quality foods, such as fruits and vegetables, have worse diet quality that children in households that are food secure. Additionally, evidence from adult studies link household FI to MASLD and liver fibrosis, and prior research of the PI has shown that exposure to household FI in early childhood was associated with a nearly 4 times increased odds of pediatric MASLD in middle childhood. Possible mechanisms linking household FI to pediatric MASLD include lower intake of fruits and vegetables, higher intake of caloric dense nutrient poor foods (e.g., sugar sweetened beverages), and less diversity of foods. Given consensus recommendations for the management of MASLD focus on lifestyle modification, i.e., diet and exercise to achieve weight loss, this proposal seeks to explore the association of household FI and pediatric MASLD disease severity and whether those effects are mediated by dietary intake. Study participants include children/adolescents with MASLD who are receiving care at UCSF's liver clinic and Weight Management for Teen and Child Health (WATCH) Clinic, a pediatric subspecialty clinic.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is now the most common type of chronic liver disease among children and adolescents in the US, with the highest burden among children from low-income families, those with obesity, and those who are Hispanic. MASLD describes a spectrum of liver injury from simple hepatic steatosis to steatohepatitis, which can progress to liver fibrosis, cirrhosis, hepatocellular carcinoma, and liver failure. MASLD is one of the leading indications for liver transplantation in adults. Emerging evidence in adults links household FI to MASLD, liver fibrosis, and mortality. FI is defined by the US Department of Agriculture (USDA) as a state in which there is "limited or uncertain availability of nutritionally adequate and safe foods or limited or uncertain ability to acquire foods in socially acceptable ways." Adults with MASLD and FI have been shown to have poor diet quality that is significantly associated with fibrosis.

Research has found that household FI is highly prevalent in families with children. Fifteen percent of U.S. households, and 30% of San Francisco households with children are food insecure, which limits the ability of these families to consistently provide healthy, high-quality food. Research has found that children living in food insecure households have worse diet quality with regard to specific food categories compared to those in food secure households. Specifically children in food insecure households consume fewer fruits and vegetables (F&V), and more SSBs. Children in households with severe FI have worse overall diet quality than those who are food secure.

Researchers, including the PI (see preliminary studies below), have found that exposure to household FI in children/adolescents is associated with pediatric MASLD. Given current consensus recommendations for the management of pediatric MASLD focus on lifestyle interventions, i.e., diet and physical activity), this project will assess the association of household FI and MASLD disease severity and whether these effects are mediated by dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents receiving care in the liver and WATCH clinics.
* Family living in California.
* Parent/guardian speaks Spanish or English.
* Child is between the ages of 6 to <17 years.
* Elevated ALT on at least 2 occasions within the past year:

  * ALT > 22 units/L for females.
  * ALT > 26 units/L for males.
* BMI for age/sex ≥ 85%.
* Alternatively, child has one elevated ALT within the past year and confirmed steatosis on imaging.
* Family does not intend to move out of California within the next year.
* Family is not already receiving EatSF SF Fruit and Vegetable Vouchers.
* Family is not participating in any other dietary education programs besides those offered by the WATCH or liver clinics.

Exclusion Criteria:

* Child has an underlying condition or medication causing their weight gain (e.g., hypothyroidism, Prader-Willi syndrome, antipsychotic medications).
* Child is on, or expected to go on, or starts on a weight loss medication (e.g., Qsymia or GLP-1 receptor agonists).
* Child has another known cause of liver disease (not including MASLD or MASH), such as:

  * Autoimmune hepatitis.
  * Wilson's disease.
  * Hepatitis A, B, or C.
  * Acute infection.
  * Genetic condition causing inflammation in the liver.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with MASLD with and without exposure to household food insecurity.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase (ALT) | 30 days
  Alanine aminotransferase (ALT)
Gamma-glutamyl transferase (GGT) | 30 days
  Gamma-glutamyl transferase (GGT)

SECONDARY OUTCOMES:
Dietary intake of fruits and vegetables | 30 days
  Dietary intake of fruit and vegetables
dietary intake of SSBs | 30 days
  Dietary intake of sugar sweetened beverages

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Maxwell, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golovaty I, Tien PC, Price JC, Sheira L, Seligman H, Weiser SD. Food Insecurity May Be an Independent Risk Factor Associated with Nonalcoholic Fatty Liver Disease among Low-Income Adults in the United States. J Nutr. 2020 Jan 1;150(1):91-98. doi: 10.1093/jn/nxz212. PMID 31504710
- [Background] Tamargo JA, Sherman KE, Campa A, Martinez SS, Li T, Hernandez J, Teeman C, Mandler RN, Chen J, Ehman RL, Baum MK. Food insecurity is associated with magnetic resonance-determined nonalcoholic fatty liver and liver fibrosis in low-income, middle-aged adults with and without HIV. Am J Clin Nutr. 2021 Mar 11;113(3):593-601. doi: 10.1093/ajcn/nqaa362. PMID 33515016
- [Background] Kardashian A, Dodge JL, Terrault NA. Food Insecurity is Associated With Mortality Among U.S. Adults With Nonalcoholic Fatty Liver Disease and Advanced Fibrosis. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2790-2799.e4. doi: 10.1016/j.cgh.2021.11.029. Epub 2021 Dec 16. PMID 34958747
- [Background] Kardashian A, Dodge JL, Terrault NA. Racial and ethnic differences in diet quality and food insecurity among adults with fatty liver and significant fibrosis: a U.S. population-based study. Aliment Pharmacol Ther. 2022 Nov;56(9):1383-1393. doi: 10.1111/apt.17219. Epub 2022 Sep 29. PMID 36173037
- [Background] Landry MJ, van den Berg AE, Asigbee FM, Vandyousefi S, Ghaddar R, Davis JN. Child-Report of Food Insecurity Is Associated with Diet Quality in Children. Nutrients. 2019 Jul 12;11(7):1574. doi: 10.3390/nu11071574. PMID 31336880
- [Background] Maxwell SL, Price JC, Perito ER, Rosenthal P, Wojcicki JM. Food insecurity is a risk factor for metabolic dysfunction-associated steatotic liver disease in Latinx children. Pediatr Obes. 2024 Jun;19(6):e13109. doi: 10.1111/ijpo.13109. Epub 2024 Mar 7. PMID 38453472